CLINICAL TRIAL: NCT00196898
Title: A National, Multicenter Study on Fibrotic Valvular Heart Disease in Patients With Parkinson´s Disease Treated With Dopamine Agonists
Brief Title: Multicenter Study on Fibrotic Valvular Heart Disease in Patients With Parkinson's Disease Treated With Dopamine Agonists
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Parkinson Study Group (GPS) (Other)
Collaborators: Competence Network on Parkinson's Disease (Other)
Responsible Party: Competence Network on Parkinson´s disease, Dr. Karla Eggert, Competence Network on Parkinson´s disease
Other Study IDs: 1.0 / 03.02.05; Grant 01 GI 0201/01 GI 0401
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-04

CONDITIONS: Heart Valve Diseases; Parkinson's Disease
Keywords: Parkinson´s disease; fibrotic valvular heart fibrosis; ergot dopamine agonists; non-ergot dopamine agonists
MeSH Terms: conditions — Heart Valve Diseases; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Fibrotic valvular heart diseases are known as rare complications of long-time therapy of Parkinson's disease with ergot-derivatives including some ergot-dopamine agonists. The aim of this study is to assess the incidence of valvular heart disease, which may be an ergot-drug agonists side-effect or an overall complication of all dopamine agonists. Incidence, prevalence and addiction of dose or intake duration are not known so far. The reversibility of the changes is unknown too. To answer these questions the present study is designed as a cross sectional study followed by a 2 year follow-up prospective cohort study.

DETAILED DESCRIPTION:
Rare incidence of pleuropulmonary and retroperitoneal fibrosis are known complications during the long-time therapy of Parkinson's disease (PD) with ergot-drug derivatives including some ergot dopamine agonists. Particularly the appearance of fibrotic valvular heart disease of Parkinson patients under Pergolide therapy caused an intense discussion about the safety of dopamine agonists at all. Single case reports of similar heart valve changes under the therapy of Bromocriptin and probably Cabergoline pointed to an effect of the whole substance class of the ergot-dopamine agonists.

Cross-Sectional Study (part I):

Within this study an initial cross-sectional analysis of the prevalence of fibrotic heart valvular disease will be done. Patients with Parkinson's disease with different exposition status will be recruited. An transthoracal echocardiographic examination (TTE) of the heart will be performed.

Exposition status:

* patients with ergot-derived dopamine agonists
* patients with non-ergot-derived dopamine agonists
* After the TTE-report the study population is divided in affected (= pathological TTE-report: fibrotic valvular heart diseases) and healthy persons (= non-pathological TTE-report: no fibrotic valvular heart diseases). The therapy with dopamine agonist will be stopped in patients with a pathological TTE-report. Instead these patients will be treated with an equivalent dose of L-Dopa with or without COMT-inhibitors. The existing therapy regime will remain in patients without pathological findings.

Longitudinal Section (part II and III):

The cross-sectional study (part I) is followed by a two year follow-up study.

Cohort I:

* patients with pathological TTE-report: fibrotic valvular heart disease
* patients without pathological TTE-report: no fibrotic valvular heart disease

Part II: Within cohort I the reversibility of fibrotic valvular heart disease will be analysed with regard to the previously taken cumulative dose of dopamine agonists.

Part III: Within cohort II there will be a prospective analysis of the (cumulative) incidence of fibrotic valvular heart disease in PD patients with different exposition status. If fibrotic valvular heart disease occurs, a patient will be changed from cohort II to cohort I.

Primary Outcome:

Cross-sectional study (part I):

* What is the prevalence of fibrotic valvular heart disease in PD patients under therapy with ergot-derived dopamine agonists and non-ergot-derived dopamine agonists?
* Is there an influence to the cumulative dose of dopamine agonists?

Longitudinal study (prospective cohort study):

* (Part II) Is fibrotic valvular heart disease under therapy of ergot-derived dopamine agonists and non-ergot-derived dopamine agonists reversible?
* (Part III) What is the (cumulative) incidence of fibrotic valvular heart disease under the therapy of ergot-derived dopamine agonists and non-ergot-derived dopamine agonists?

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of Morbus Parkinson
* Written informed consent

Exclusion Criteria:

* Patients with a history of carcinoid syndrome
* Patients with a history of post-inflammatory (rheumatic), degenerative (calcified) or ischaemic coronary heart or valvular heart disease
* Previous medication with ergot-derived drugs (eg. Methysergide, Ergotamine) except dopamine receptor agonists or anorectic drugs (eg. Fenfluramine, Dexfenfluramine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD Patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-03; Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Oertel, Prof. Dr., Study Chair — Universitätsklinikum Marburg und Gießen
Locations (1):
- Universitätsklinikum Marburg und Gießen, Neurologische Klinik, Marburg, Hesse, Germany

REFERENCES:
- See also: Homepage Competence Network on Parkinson's disease sponsored by the German government — http://www.kompetenznetz-parkinson.de